CLINICAL TRIAL: NCT07039838
Title: Cardiac Computed Tomography Based 3-D Printing for Optimized Coronary Artery Bypass Graft Surgery
Acronym: 3DCABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jesper James Linde (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jesper James Linde, Consulting Cardiologist, Associate Professor, Head of Cardiac Imaging Unit at the Department of Cardiology, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-24070405; H-24070405 (Other: The Committees on Health Research Ethics in the Capital Region of Denmark)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Coronary Arterial Disease (CAD); Bypass Graft Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Will undergo CABG as per usual clinical practice
- 3D-print guided CABG (Experimental): Will have a CT-based 3D-print of the coronary arteries marked with the optimal graft insertion points to be used during CABG
  Interventions: Diagnostic Test: 3D print of coronary arteries

INTERVENTIONS:
Diagnostic Test: 3D print of coronary arteries — Based on a pre-surgical cardiac CT the optimal graft insertions points on the target coronary arteries wil be marked and a patient-specific model of the coronary arteries will be 3D-printed and sterialized to be available during CABG to guide the placement of the distal graft anastomosis.
  Arms: 3D-print guided CABG

SUMMARY:
Coronary artery bypass graft surgery (CABG) is a preferred surgical treatment in patients with widespread coronary artery disease. However, studies have shown that up to one third of patients will have closure of at least one bypass graft (graft failure) after one year, which has prognostic implications. Since graft failure can partly be due to inappropriate placement of the distal graft anastomosis, there is a need to develop new surgical methods to ensure optimal placement of the grafts. Three-dimensional (3D) printing is a technique developed to transform digital objects into physical models. The method is widely used in orthopedic surgery and maxillofacial surgery, but has also gained interests in cardiology, and has proved usefull in the preparation for invasive interventions or surgery in patients with complicated anatomy, including congenital heart disease.

The purpose of the study is to investigate, if a surgical strategy, based on a preoperative cardiac CT, including a patient-specific printed 3-D model of the coronary vessels, marked with optimal bypass graft insertion points, can reduce graft failure, assessed by a control cardiac CT examination performed 12 months after surgery. The hypothesis is that 3-D printing of coronary vessels determined from invasive coronary angiography and cardiac CT prior to CABG reduces graft failure 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Indication for CABG (with or without valve-surgery), determined by heart team conference. The revascularization plan must include further grafting in addition LIMA to LAD.

Exclusion Criteria:

* Age <18 years

  * Permanent atrial fibrillation
  * Renal failure (eGRF < 30)
  * Known allergy to contrast material
  * Pregnant and/or breastfeeding
  * Indication for acute CABG
  * Patients who cannot tolerate premedication with nitroglycerin and beta blocker (including LVEF<40%). This applies only to the pre-operative CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Graft failure | From surgery to the control cardiac CT performed at 12 months
  Difference in the proportion of grafts with graft failure 12 months after surgery. Graft failure is defined as: 1) graft occlusion 2) graft stenosis >50% 3) Graft anastomosis is placed on wrong vessels or proximal to the stenosis 4) String sign (radialis grafts)

SECONDARY OUTCOMES:
Graft failure at a patient level | From surgery to the control cardiac CT performed at 12 months
  Difference in the proportion of patients with graft failure at 12 months
Occluded grafts | From surgery to the control cardiac CT at 12 months
  Difference in number of occluded grafts at 12 months (graft level and patient level)
Graft stenosis | From surgery to the control cardiac CT at 12 months
  Difference in proportion of graft stenosis at 12 months (graft level and patient level)
Grafts placed on wrong vessels or proximal to coronary stenosis | From surgery to the control cardiac CT at 12 months
  Difference in the number of grafts placed on wrong vessels or proximal to coronary stenosis (graft level and patient level)
Acute myocardial infarction or new revascularization | From surgery to the control cardiac CT at 12 months
  Acute myocardial infarction or renewed revascularization at 12 months.
Hospitalization for chest pain, acute coronary disease, heart failure or death | From surgery to the control cardiac CT at 12 months
  Hospitalization with chest pain, acute coronary disease, heart failure or death at 12 months

OTHER OUTCOMES:
Myocardial perfusion | From surgery to the control Cardiac CT performed at 12 months
  Difference in myocardial perfusion assessed by cardiac CT scan at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
We do not have approval to share patient data with other researchers